CLINICAL TRIAL: NCT02859311
Title: A Pilot Feasibility Study in Recovered Heart Failure
Acronym: TRED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015CD007B
Record Dates: First submitted 2016-04-14; First posted 2016-08-09 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Heart Failure
Keywords: Recovery
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Withdrawal of therapy (Experimental): Gradual, supervised withdrawal of medical therapy over 4-16 weeks
  Interventions: Drug: Withdrawal of therapy
- Control (No Intervention): Continuation of usually prescribed pharmacological therapy

INTERVENTIONS:
Drug: Withdrawal of therapy — Withdrawal of heart failure therapies (angiotensin converting enzyme inhibitors, angiotensin receptor blockers, beta-blockers, mineralocorticoid receptor antagonists and loop diuretics)
  Arms: Withdrawal of therapy

SUMMARY:
One third of patients diagnosed with heart failure demonstrate left ventricular reverse remodelling and recovery of cardiac function following a period of medical therapy. These patients have an excellent long-term prognosis. Whether they need to remain on long-term medical therapy is not clear. The investigators will investigate the safety of therapy withdrawal in patients with a previous diagnosis of heart failure and recovered cardiac function, in a randomised controlled trial.

DETAILED DESCRIPTION:
Patients with a previous diagnosis of heart failure, who have recovered cardiac function, without symptoms, normal serum biomarker concentrations and who are currently still taking heart failure medications, will be recruited. Participants will be randomised to withdrawal of therapy and control arms and will undergo imaging investigations and cardiopulmonary exercise tests at baseline along with serum biomarker tests. Those participants randomised to withdrawal of therapy will have a gradual, supervised reduction of medications. If, at anytime, there are signs of recurring heart failure, medications will be restarted. Participants in the control arm will continue their medical therapy as usual.

Participants will be followed up with further biomarker testing, cardiopulmonary exercise testing and imaging investigations at 6 months.

The primary end-point will be a relapse in heart failure, defined by adverse remodelling, increase in left ventricular size, rise in serum biomarkers or clinical evidence of heart failure as judged by the clinical team.

ELIGIBILITY:
Inclusion Criteria:

1. Have an index diagnosis of heart failure confirmed by 2 independent operators based on clinical details.
2. Be currently taking at least 1 of the following medications loop diuretic, betablocker, angiotension converting enzyme inhibitor/angiotensin receptor blocker and mineralocorticoid receptor antagonist.
3. Have demonstrated evidence of left ventricular reverse remodelling following the initial diagnosis with subsequent improvement in ejection fraction to >50% and normalisation of left ventricular (LV) volumes.
4. Have no symptoms of heart failure (NYHA Class 1).
5. Low plasma NTproBNP.

Exclusion Criteria:

1. Uncontrolled hypertension.
2. More than moderate valvular disease.
3. Estimated glomerular filtration rate <30mls/min.
4. Atrial/supraventricular/ventricular arrhythmia requiring beta-blockade.
5. Pregnancy.
6. Unstable angina.
7. Age <16 years

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Heart failure relapse | 6 months
  Defined by one of the following: 1) A reduction in left ventricular ejection fraction; 2) An increase in left ventricular size; 3) An increase in serum biomarker concentration from baseline; 4) Clinical evidence of heart failure

SECONDARY OUTCOMES:
Cardiopulmonary exercise testing with peak oxygen consumption | 6 months
  Change in peak oxygen consumption between baseline and follow-up test
Quality of life | 6 months
  Patient questionnaires - Kansas City Cardiomyopathy Questionnaire and Heart Failure Symptom Questionnaire (symptom scores are calculated on the basis of the participants' answers to the questionnaires)
Major adverse cardiovascular events (MACE) - safety end-point | 6 months
  MACE - unplanned cardiovascular (CV) hospitalisation, CV mortality and major adverse CV events (non-fatal myocardial infarction and non-fatal cerebrovascular accident)
Percentage of participants with new and sustained arrhythmias | 6 months
  New and sustained arrhythmias diagnosed during follow-up
Increase in left atrial volume as measured on cardiovascular magnetic resonance (CMR) | 6 months
  Increase in left atrial volume as measured on CMR (in millilitres)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Prasad, MD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Halliday BP, Vazir A, Owen R, Gregson J, Wassall R, Lota AS, Khalique Z, Tayal U, Jones RE, Hammersley D, Pantazis A, Baksi AJ, Rosen S, Pennell DJ, Cowie MR, Cleland JGF, Prasad SK. Heart Rate as a Marker of Relapse During Withdrawal of Therapy in Recovered Dilated Cardiomyopathy. JACC Heart Fail. 2021 Jul;9(7):509-517. doi: 10.1016/j.jchf.2021.03.010. Epub 2021 Jun 9. PMID 34119469
- [Derived] Halliday BP, Wassall R, Lota AS, Khalique Z, Gregson J, Newsome S, Jackson R, Rahneva T, Wage R, Smith G, Venneri L, Tayal U, Auger D, Midwinter W, Whiffin N, Rajani R, Dungu JN, Pantazis A, Cook SA, Ware JS, Baksi AJ, Pennell DJ, Rosen SD, Cowie MR, Cleland JGF, Prasad SK. Withdrawal of pharmacological treatment for heart failure in patients with recovered dilated cardiomyopathy (TRED-HF): an open-label, pilot, randomised trial. Lancet. 2019 Jan 5;393(10166):61-73. doi: 10.1016/S0140-6736(18)32484-X. Epub 2018 Nov 11. PMID 30429050